CLINICAL TRIAL: NCT07103395
Title: A Phase II Study Evaluating Neoadjuvant Chemotherapy, Concurrent Chemoradiotherapy Combined With Dual Immune Checkpoint Blockade (PD-1/CTLA-4) in Patients With Locally Advanced Non-Small Cell Lung Cancer
Brief Title: A Study Evaluating Neoadjuvant Chemotherapy, Concurrent Chemoradiotherapy Combined With Dual Immune Checkpoint Blockade in Patients With Locally Advanced Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-10135
Record Dates: First submitted 2025-07-16; First posted 2025-08-05 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer (NSCLC)
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The study group (Experimental): Patients will receive neoadjuvant chemotherapy combined with iparomlimab and tuvonralimab and thymosin alpha 1, followed by concurrent chemoradiotherapy, and finally consolidation therapy with iparomlimab and tuvonralimab and thymosin alpha 1.
  Interventions: Drug: Neoadjuvant therapy; Radiation: Radiotherapy; Drug: Consolidative therapy

INTERVENTIONS:
Drug: Neoadjuvant therapy — The neoadjuvant regimen prior to radiotherapy consists of albumin-bound paclitaxel/pemetrexed, cisplatin, Bevacizumab, iparomlimab and tuvonralimab, and thymosin alpha 1.
Radiation: Radiotherapy — Definitive dose of hypofractionated radiotherapy was delivered to patients, with concurrent chemotherapy and surufatinib.
Drug: Consolidative therapy — Consolidation therapy consists of iparomlimab and tuvonralimab, surufatinib and thymosin alpha 1, for a total duration of 1 year.

SUMMARY:
This study will enroll patients with locally advanced non-small cell lung cancer (NSCLC). Patients will receive neoadjuvant chemotherapy combined with dual immune checkpoint blockade (PD-1/CTLA-4), bevacizumab and thymosin alpha 1, followed by concurrent chemoradiotherapy, and finally consolidation therapy with dual immune checkpoint blockade (PD-1/CTLA-4), surufatinib and thymosin alpha 1. The study aims to evaluate the efficacy and safety of this treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 to 75 years or older;
* Patients must have histologically or cytologically confirmed locally advanced, unresectable (Stage III) non-small cell lung cancer (NSCLC);
* EGFR, ALK, and ROS1 wild-type;
* No prior chemotherapy, radiotherapy, surgery, targeted therapy, or immunotherapy;
* Expected survival ≥ 12 weeks;
* WHO Performance Status (PS) score of 0 or 1;
* Female subjects must not be breastfeeding;
* Women of childbearing potential (WOCBP) must agree to use contraception during the study treatment and for 5 months after the last dose of study drug (i.e., 30 days [one ovulation cycle] plus approximately five half-lives of the study drug);
* Adequate organ and bone marrow function as defined by the following criteria:
* Forced Expiratory Volume in 1 second (FEV1) ≥ 800 mL;
* Absolute neutrophil count ≥ 1.5 × 10⁹/L;
* Platelets ≥ 100 × 10⁹/L;
* Hemoglobin ≥ 9.0 g/dL;
* Creatinine clearance ≥ 50 mL/min as calculated by the Cockcroft-Gault formula (Cockcroft and Gault, 1976);
* Serum bilirubin ≤ 1.5 × upper limit of normal (ULN);
* AST and ALT ≤ 2.5 × ULN.

Exclusion Criteria:

1. Exclusion criteria for enrolment for neoadjuvant therapy. Patients should not enter the study if any of the following exclusion criteria are fulfilled:

   * Concurrent enrolment in another clinical study, unless it is an observational(non-interventional) clinical study;
   * Mixed small cell and non-small cell lung cancer histology;
   * Prior use of anti-PD-1, anti-PD-L1, or anti-CTLA4 antibodies;
   * Recent major surgery within 4 weeks prior to entry into the study (excluding the placement of vascular access;
   * Active or prior documented autoimmune disease within the past 2 years;
   * Active or prior documented inflammatory bowel disease (eg. Crohn's disease, ulcerative colitis);
   * History of primary immunodeficiency;
   * History of organ transplant that requires therapeutic immunosuppression;
   * Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any patient known to have hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the patient to give written informed consent;
   * Known history of tuberculosis;
   * History of another primary malignancy within 5 years prior to starting treatment, except for adequately treated basal or squamous cell carcinoma of the skin or cancer of the cervix in situ and the disease under study;
   * Female patients who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control.
2. Exclusion criteria for concurrent chemoradiation following neoadjuvant therapy. Patients should not enter the concurrent chemoradiation phase if any of the following exclusion criteria are fulfilled:

   * Patients who develop distant metastasis;
   * Patients who develop locoregional disease progression and the irradiation dose of normal tissue will exceed the limit.
   * World Health Organization (WHO) Performance Status of 2-4;
   * Inadequate organ and marrow function as defined below:

     * Forced expiratory volume in 1 second (FEV1) <800ml
     * Absolute neutrophil count <1.5 x 109/L (1500 per mm3)
     * Platelets <100 x 109/L (100,000 per mm3)
     * Haemoglobin<9.0 g/dL (5.59 mmol/L)
     * Serum creatinine CL <50 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976)
     * Serum bilirubin >1.5 x upper limit of normal (ULN).
     * Aspartate Transaminase(AST) and Alanine Transaminase(ALT) >2.5 x ULN.
3. Further exclusion criteria for consolidation therapy. Patients should not enter the consolidation therapy if any of the following exclusion criteria are fulfilled:

   * Patients who have progressed whilst definitive platinum based, concurrent chemoradiation therapy;
   * Current or prior use of immunosuppressive medication within 28 days before the first dose of Iparomlimab and tuvonralimab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Systemic steroid administration required to manage toxicities arising from radiation therapy delivered as part of the chemoradiation therapy for locally advanced NSCLC is allowed.
   * Any unresolved toxicity CTCAE >Grade 2 from the prior chemoradiation therapy will be excluded from randomization;
   * Patients with Grade ≥2 pneumonitis from prior chemoradiation therapy will be excluded from randomization;
   * Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE>Grade 1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2029-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2-year
  PFS measures the time from the start date of treatment to disease progression, death from any cause or last follow up if alive.

SECONDARY OUTCOMES:
Objective response rate | 2 month after treatment
Overall survival | 2-year
  OS measures the time from the start date of treatment to death from any cause or last follow up if alive.
Treatment-related toxicity | through study completion, an average of 18 months
  Treatment-related toxicities were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) 5.0 toxicity

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Danielli R, Cisternino F, Giannarelli D, Calabro L, Camerini R, Savelli V, Bova G, Dragonetti R, Di Giacomo AM, Altomonte M, Maio M. Long-term follow up of metastatic melanoma patients treated with Thymosin alpha-1: investigating immune checkpoints synergy. Expert Opin Biol Ther. 2018 Jul;18(sup1):77-83. doi: 10.1080/14712598.2018.1494717. PMID 30063847
- [Background] Garaci E, Pica F, Rasi G, Favalli C. Thymosin alpha 1 in the treatment of cancer: from basic research to clinical application. Int J Immunopharmacol. 2000 Dec;22(12):1067-76. doi: 10.1016/s0192-0561(00)00075-8. PMID 11137613
- [Background] Garaci E, Pica F, Serafino A, Balestrieri E, Matteucci C, Moroni G, Sorrentino R, Zonfrillo M, Pierimarchi P, Sinibaldi-Vallebona P. Thymosin alpha1 and cancer: action on immune effector and tumor target cells. Ann N Y Acad Sci. 2012 Oct;1269:26-33. doi: 10.1111/j.1749-6632.2012.06697.x. PMID 23045967
- [Background] Provencio M, Nadal E, Insa A, Garcia-Campelo MR, Casal-Rubio J, Domine M, Majem M, Rodriguez-Abreu D, Martinez-Marti A, De Castro Carpeno J, Cobo M, Lopez Vivanco G, Del Barco E, Bernabe Caro R, Vinolas N, Barneto Aranda I, Viteri S, Pereira E, Royuela A, Casarrubios M, Salas Anton C, Parra ER, Wistuba I, Calvo V, Laza-Briviesca R, Romero A, Massuti B, Cruz-Bermudez A. Neoadjuvant chemotherapy and nivolumab in resectable non-small-cell lung cancer (NADIM): an open-label, multicentre, single-arm, phase 2 trial. Lancet Oncol. 2020 Nov;21(11):1413-1422. doi: 10.1016/S1470-2045(20)30453-8. Epub 2020 Sep 24. PMID 32979984
- [Background] Huang Y, Yang Y, Zhao Y, Zhao H, Zhou N, Zhang Y, Chen L, Zhou T, Chen G, Wu T, Lu L, Xue S, Kang X, Zhang L, Fang W. QL1706 (anti-PD-1 IgG4/CTLA-4 antibody) plus chemotherapy with or without bevacizumab in advanced non-small cell lung cancer: a multi-cohort, phase II study. Signal Transduct Target Ther. 2024 Jan 29;9(1):23. doi: 10.1038/s41392-023-01731-x. PMID 38282003
- [Background] Cheng W, Kang K, Zhao A, Wu Y. Dual blockade immunotherapy targeting PD-1/PD-L1 and CTLA-4 in lung cancer. J Hematol Oncol. 2024 Jul 27;17(1):54. doi: 10.1186/s13045-024-01581-2. PMID 39068460